CLINICAL TRIAL: NCT04748276
Title: Tracking Response to Antidepressants in Advance of Investigational Trials
Acronym: TRAIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Adams Clinical (Network)
Responsible Party: Sponsor
Other Study IDs: TRAIT-MDD-107
Record Dates: First submitted 2021-02-07; First posted 2021-02-10 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: FDA-approved selective-serotonin reuptake inhibitors (SSRIs) and selective-norepinephrine reuptake inhibitors (SNRIs) — Protocol-approved antidepressant treatments (ADT) will be prescribed in accordance with standard of care, whenever possible following dosing recommendations within the Study Formulary and Prescribing Guidelines (Sertraline 100 mg/day; Citalopram 20 mg/day; Escitalopram 10 mg/day; Fluoxetine 20 mg/day; Paroxetine 20 mg/day; Duloxetine 60 mg/day; Buproprion 300 mg/day; Desvenlafaxine 50 mg/day; Venlafaxine 150 mg/day). ADTs may be up or down-tapered as necessary.

SUMMARY:
TRAIT is an open-label observational study to evaluate treatment response to selective-serotonin reuptake inhibitors (SSRIs) and selective-norepinephrine reuptake inhibitors (SNRIs) among individuals meeting criteria for Major Depressive Disorder (MDD) and seeking enrollment in investigational trials.

ELIGIBILITY:
Inclusion Criteria:

* Participant has signed an ICF prior to any study-specific procedures being performed.
* Participant is male or female of age ≥ 18 years old.
* Participant has a diagnosis of MDD as confirmed by the MINI semi-structured diagnostic interview and ≥ 14 HAM-D total score.
* Participant is in good physical health and, in the opinion of the investigator, is a suitable candidate for treatment with an ADT.

Exclusion Criteria:

* Participant is pregnant, breast-feeding, or planning to become pregnant.
* A history or presence of a clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, or neurologic abnormality, which in the opinion of the investigator may impact participant safety or study results.
* Participant has a history of any psychiatric condition other than MDD, which in the opinion of the investigator is primary, or any other psychiatric or neurologic disorder or symptom that could pose undue risk to the participant or compromise the study.
* Any participant who represents an acute suicidal risk in the opinion of the investigator.
* Moderate or severe substance use disorder within 90 days prior to screen, according to DSM-5 criteria that in the opinion of the investigator could pose undue risk to the participant, or compromise the study.
* Any condition that, in the opinion of the investigator, makes the participant unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who currently meet the Diagnostic and Statistical Manual - Version 5 (DSM-5) criteria for Major Depressive Disorder and are seeking enrollment in an industry-sponsored clinical trial of a second- or third-line antidepressant.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Inventory - 17 item (HAM-D) total score in response to a treatment cycle from Baseline/Day 0 to the end of a 6-week treatment cycle. | Up to 33 weeks

SECONDARY OUTCOMES:
Failure to respond to 1, 2, or 3+ ADT treatment cycles, as defined as < 25% change in HAM-D total score from study Baseline/Day 0 to Day 42 of the participant's 1st, 2nd, or 3rd+ treatment cycles. | Up to 33 weeks
Partial response to 1, 2, or 3+ ADT treatment cycles, as defined as ≥ 25% to < 50% change in HAM-D total score from study Baseline/Day 0 to Day 42 of the participant's 1st, 2nd, or 3rd+ treatment cycles. | Up to 33 weeks
Total number of treatment cycles required to reach ADT response, as defined as ≥ 50% reduction in HAM-D score from Baseline/Day 0 to Day 42 of each treatment cycle. | Up to 33 weeks

OTHER OUTCOMES:
Presence of and change in anxiety symptoms as assessed by the MDD with Anxious Distress subscale of the Mini-International Neuropsychiatric Inventory (MINI), and self-report on the Beck Anxiety Inventory (BAI). | Up to 33 weeks
Presence of and change in sleep-related disturbance as assessed by the self-reported Insomnia Severity Index (ISI). | Up to 33 weeks
Presence of and change in anger symptoms as assessed by the self-reported Massachusetts General Hospital Anger Attacks Questionnaire (MGH AAQ), and the self-reported Concise Associated Symptoms Tracking Scale (CAST-SR). | Up to 33 weeks
Presence of and change in depression-/treatment- related sexual dysfunction as assessed by the self-reported Change in Sexual Functioning Questionnaire (CSFQ). | Up to 33 weeks
Presence of and change in functional impairment as assessed by the Sheehan Disability Scale, Inventory of Depressive Symptomology, Short Form Survey Instruments, Patient Global Impressions, and the Clinical Global Impression scale. | Up to 33 weeks
Presence of and change in pain conditions as assessed by the self-reported Brief Pain Inventory, Short Form (BPI-SF) and Visual Analog Scale - Pain (VAS-PAIN). | Up to 33 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Ellickson, PhD, Principal Investigator — Adams Clinical
Locations (1):
- Adams Clinical, Watertown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided